CLINICAL TRIAL: NCT03438656
Title: Targeted Intervention for Adolescents Following Child Maltreatment: Examining Neural and Behavioral Mechanisms Within the Positive Valence System
Brief Title: Activating and Connecting Teens (ACT) Study
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Jenness, Acting Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002283; K23MH112872 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-20 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: Depression; Childhood adversity; Behavioral Activation; Reward Processing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation Arm (Experimental): See treatment description for information on Behavioral Activation. Participants will receive 12 weekly sessions of Behavioral Activation.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — The Adolescent Behavioral Activation Program (ABAP) will be used as the BA protocol. ABAP was developed and validated by McCauley, Dimidjian et al. to adapt BA to adolescents. ABAP is a 12-week protocol that utilizes an idiographic approach to foster rewarding experiences, effective problem solving, and goal attainment, and decrease avoidance, barriers to activation, and depressive rumination that may be contributing to depression severity and maintenance.

SUMMARY:
National data indicate over 650,000 children and adolescents are exposed to physical, sexual, or emotional abuse or physical or emotional neglect each year. Moreover, youth with a history of childhood maltreatment (CM) are at least twice as likely to develop depression and are at substantial risk for nonresponse to current best practice depression interventions (i.e., cognitive behavioral therapy and antidepressants) compared to non-maltreated peers. Research suggests that CM increases risk for depression through disruptions in the positive valence system, such as reward processing, and Behavioral Activation (BA) may be an alternative depression intervention that targets these deficits. This proposal will examine whether BA intervention reduces depression and anhedonia in a sample of depressed adolescents, aged 13-18, with variable histories of CM exposure (BA Group). A total of 30 depressed adolescents will be recruited to undergo a 12-week course of BA. All participants will undergo clinical assessment to measure depression symptoms and anhedonia at baseline (Week 0) and post- (Week 12) treatment.

ELIGIBILITY:
Inclusion Criteria Behavioral Activation Group:

- current diagnosis of clinical depression (minor or major) will be recruited as study participants in the Behavioral Activation (BA) Group

Exclusion Criteria:

* IQ < 80;
* non-English speaking youth or parent;
* current PTSD diagnosis;
* lifetime history of a developmental (e.g., autism), neurological (e.g., epilepsy), psychotic, bipolar, or substance disorder;
* current psychiatric (e.g., antidepressants) or other mood altering medication (e.g., steroids) other than AD/HD medication;
* requiring a higher level of care (i.e., inpatient hospitalization) due to suicidality or other mental or physical health related problem.
* Any youths who are currently being maltreated will not be enrolled to ensure that participants do not have active safety concerns.
* Full course of other evidence-based depression intervention

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Jenness, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We did not assign to groups. This was a single-arm, open pilot trial
Period: Overall Study
Arm/Group | Behavioral Activation Arm
Started | 32
Completed | 30
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Activation Arm
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.88 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 12
  More than one race | 9
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Changes in depression symptoms will be measured with self-report on the Patient Health Questionnaire-9 (PHQ-9). Total score will be reported with a range of 0 to 27 with higher scores indicating greater symptoms of depression. Higher symptoms of depression are considered a worse outcome.
  units on a scale | 13.94 (6.51)
Childhood Trauma Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Childhood Trauma Questionnaire (CTQ) measures lifetime experiences of sexual, physical, and emotional abuse as well as emotional neglect. The total score ranges from 5 to 125 with higher scores indicating more experiences of abuse or neglect.
  units on a scale | 40.63 (9.00)
Anhedonia [Mean (Standard Deviation); unit: units on a scale] — Changes in feelings of loss of pleasure and interest (i.e., Anhedonia) will be measured via self-report on the Behavioral Activation for Depression Scale (BADS) total score. The range on the BADS is 0 to 150, with higher scores representing less activation. Higher scores are considered a worse outcome on this measure.
  units on a scale | 73.53 (22.18)

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Changes in depression symptoms will be measured with self-report on the Patient Health Questionnaire-9 (PHQ-9). Total score will be reported with a range of 0 to 27 with higher scores indicating greater symptoms of depression. Higher symptoms of depression are considered a worse outcome.
Time Frame: Week 12 (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Arm
Number analyzed (Participants) | 32
score on a scale | 9.63 (5.49)

2. Primary Outcome: Anhedonia/Activation
Description: Changes in feelings of loss of pleasure and interest (i.e., Anhedonia) will be measured via self-report on the Behavioral Activation for Depression Scale (BADS) total score. The range on the BADS is 0 to 150, with higher scores representing less activation. Higher scores are considered a worse outcome on this measure.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation Arm
Number analyzed (Participants) | 32
score on a scale | 61.80 (22.19)

3. Other Pre Specified Outcome: Anxiety
Description: Changes in anxiety symptoms and diagnoses with diagnostic interviews and self-report (SCARED).
Time Frame: Symptoms will be measured at baseline, post-treatment, and 3-month follow-up.
Reporting Status: Not Posted, anticipated posting 2024-03

4. Other Pre Specified Outcome: Behavioral Problems
Description: Changes in commonly co-morbid behavioral problems with depression (i.e., attention deficit/hyperactivity disorder, conduct problems, oppositionality) and diagnoses will be measured.
Time Frame: Pre- (Week 0) and post-treatment (Week 12)
Reporting Status: Not Posted, anticipated posting 2024-03

5. Other Pre Specified Outcome: Hopelessness
Description: Changes in feelings of hopelessness (i.e., feeling like nothing is good, everything is bad, nothing can change it) will be measured by self-report.
Time Frame: Pre- (Week 0) and post-treatment (Week 12)
Reporting Status: Not Posted, anticipated posting 2024-03

6. Other Pre Specified Outcome: Suicidality
Description: Changes in suicidal ideation, plans, and behaviors and self-harm thoughts and behaviors will be measured on a semi-structured interview and self-report.
Time Frame: Weekly throughout treatment (Weeks 0-12) and at a 3-month follow-up (24 Week)
Reporting Status: Not Posted, anticipated posting 2024-03

7. Other Pre Specified Outcome: Ecological Momentary Assessment (EMA)
Description: Changes in self-reported activity engagement and mood will be delivered through a mobile application.
Time Frame: Questionnaires delivered 3x/day, 2 days/week from Weeks 0 to 12
Reporting Status: Not Posted, anticipated posting 2024-03

ADVERSE EVENTS:
Time Frame: Adverse events were measured across 6-months.
Arm/Group | Behavioral Activation Arm
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03438656/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03438656/ICF_001.pdf